CLINICAL TRIAL: NCT03196713
Title: Quality and Efficacy of Early Intensive Autism Intervention: a Matter of Trust, Knowledge, and Supervision?
Brief Title: Early Intervention, Supervision, Quality and Outcome in ASD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Sven Bölte, Head of Neuropsychiary Division, director of KIND, Professor, PhD, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: EIBI Quality
Record Dates: First submitted 2017-06-20; First posted 2017-06-23 (Actual); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Autism Spectrum Disorder
Keywords: Allegiance; Knowledge; Supervision; Early intervention; Autism
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder | interventions — Applied Behavior Analysis

STUDY DESIGN:
Intervention Model Description: Pragmatic RCT
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tailored supervision (Other)
  Interventions: Behavioral: Early Intensive Behavioral Intervention
- Regular supervision (Other)
  Interventions: Behavioral: Early Intensive Behavioral Intervention

INTERVENTIONS:
Behavioral: Early Intensive Behavioral Intervention
  Other Names: Applied Behavior Analysis

SUMMARY:
The objective of this study is to examine the significance of knowledge of autism spectrum disorder (ASD), and early intensive behavioral intervention, as well as trust in EIBI, adequate assessment of EIBI quality, and EIBI supervision on EIBI intervention outcome in ASD.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ASD (ICD-10), ongoing EIBI program

Exclusion Criteria:

-

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2013-04-01 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2017-10-27 (Actual)

PRIMARY OUTCOMES:
York Measure of Quality of Behavioural Intensive Intervention (YMQI) | Change is assessed from baseline (probe 1) to probe 2 (2-3 months), and probe 3 (4-6 months)

SECONDARY OUTCOMES:
Vineland Adaptive Behavior Scales (VABS) | Change is assessed from baseline (probe 1) to probe 2 (2-3 months), and probe 3 (4-6 months)
Social Responsiveness Scale (SRS) | Change is assessed from baseline (probe 1) to probe 2 (2-3 months), and probe 3 (4-6 months)

CONTACTS AND LOCATIONS:
Overall Officials: Sven Bolte, Prof, PhD, Principal Investigator — Karolinska Institutet, KBH, KIND
Locations (1):
- KIND, CAP Research Center, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Langh U, Cauvet E, Hammar M, Bolte S. Cross-Cultural Validation of the York Measure of Quality of Intensive Behavioral Intervention. Behav Modif. 2017 Nov;41(6):808-828. doi: 10.1177/0145445517719397. Epub 2017 Jul 9. PMID 28691542
- [Background] Langh U, Hammar M, Klintwall L, Bolte S. Allegiance and knowledge levels of professionals working with early intensive behavioural intervention in autism. Early Interv Psychiatry. 2017 Oct;11(5):444-450. doi: 10.1111/eip.12335. Epub 2016 Apr 6. PMID 27060473